CLINICAL TRIAL: NCT02414750
Title: A Phase II, Open-Label, Multicenter Study of Vemurafenib Plus Cobimetinib (GDC-0973) in Unresectable Stage IIIc or Stage IV Melanoma; Response Monitoring and Resistance Prediction With Positron Emission Tomography and Tumor Characteristics
Brief Title: Vemurafenib Plus Cobimetinib in Metastatic Melanoma
Acronym: REPOSIT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual and changing treatment landscape
Sponsor: Netherlands Working Group on Immunotherapy of Oncology (Other)
Collaborators: Hoffmann-La Roche (Industry); Amsterdam UMC, location VUmc (Other); The Netherlands Cancer Institute (Other)
Responsible Party: Principal Investigator, A.J.M. van den Eertwegh, Medical Oncologist, Netherlands Working Group on Immunotherapy of Oncology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: M14REP
Record Dates: First submitted 2015-02-11; First posted 2015-04-13 (Estimated); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Metastatic Melanoma
Keywords: Vemurafenib/cobimetinib (GDC-0973); Melanoma; Positron Emission Tomography; Tumor Characteristics; Response monitoring; Resistance prediction; molecular targeted therapy
MeSH Terms: conditions — Melanoma | interventions — Vemurafenib; cobimetinib; Positron-Emission Tomography; Biopsy; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with BRAF/MEK inhibitor (Experimental): Treatment with vemurafenib 2dd 960 mg 28/28 plus cobimetinib 1dd 60 mg 21/28. During treatment patient will undergo PET scanning with FLT and FDG, to compare both types of PET scanning.
  During the study biopsies and blood will be taken from the patients.
  Interventions: Drug: Vemurafenib plus cobimetinib; Device: Positron Emission Tomography; Procedure: Tissue sampling; Procedure: Blood sampling

INTERVENTIONS:
Drug: Vemurafenib plus cobimetinib — Molecular targeted therapy for BRAF mutated advanced melanoma patients
  Other Names: Zelboraf plus GDC-0973
Device: Positron Emission Tomography — Patient will need to undergo FDG and FLT PET scanning before and during treatment, and at time of progression
Procedure: Tissue sampling — Before and during treatment and at time of progression patients will undergo tissue sampling of a melanoma lesion
  Other Names: Biopsy
Procedure: Blood sampling — Before and during treatment and at time of progression patients will undergo blood sampling

SUMMARY:
This is a single arm explorative phase II clinical trial in 90 subjects with advanced stage melanoma harbouring a BRAFV600 mutation. PET imaging and molecular diagnostics are combined in order to monitor response to treatment with vemurafenib plus cobimetinib, examine development of resistance and correlate changes in metabolic/proliferative activity with extend of target inhibition.

DETAILED DESCRIPTION:
Molecular targeted therapy with BRAF inhibitor vemurafenib is now currently used as first line treatment for patients with unresectable stage IIIc or metastatic melanoma harboring the BRAFV600 mutation, which is present in about 50% of melanoma patients. Despite the improvement in Progression Free Survival (PFS) en Overall Survival (OS) compared to dacabarzine, acquired resistance that develops in virtually all patients treated with vemurafenib is a great concern.

Combining a BRAF inhibitor with a MEK inhibitor that targets the MAPK pathway further downstream, however, may overcome acquired resistance to BRAF inhibition and recent studies in which both MEK inhibitors and BRAF inhibitors are combined as monotherapy seem promising.

In a phase IB trial preliminary efficacy of vemurafenib with cobimetinib (GDC-0973), a highly selective inhibitor of MEK1 seems encouraging with an initial response rate of 85% and currently a phase III study of vemurafenib versus vemurafenib plus cobimetinib in BRAFV600 mutation positive patients with advanced stage melanoma is underway. It is expected that in the near future combined BRAF and MEK inhibition will be standard of care for patients with BRAFV600 mutated metastatic melanoma.

Diagnostic CT cannot assess reduction in tumor size within days after the initiation of therapy and anatomic size does not provide information about the development of therapy response or resistance at a molecular level. It has been clearly demonstrated that alterations in metabolism occur earlier than anatomical size reduction after the initiation of therapy. Molecular imaging with PET visualizes metabolic activity in tumors and is a sensitive method to detect alterations in cell metabolism, even shortly after the start of therapy. 18F-Fluorodeoxyglucose (18F-FDG) is used to visualize glucose metabolism, whereas 18F-Fluoro-3'-deoxy-3'L-fluorothymidine (18F-FLT) is used to visualize proliferation. In preclinical mouse models 18F-FLT appears to predict response or resistance to therapy better than 18F-FDG. However, so far only 18F-FDG PET has been used to monitor response to vemurafenib in some BRAFV600 mutated metastatic melanoma patients, showing a rapid decline of 18F-FDG within 2 weeks following treatment. Preclinical studies and the observation that melanoma is a highly proliferative malignancy in most patients suggest that 18F-FLT might be the radiopharmaceutical of first choice in this setting.

By detecting these metabolic alterations, responders might be distinguished from non-responders at an earlier phase compared with anatomical imaging with CT. This way, unnecessary expensive treatment of combined BRAF/MEK-inhibitor therapy and its side effects can be prevented in patients who will not benefit from this therapy. Furthermore, the level of decline in metabolic activity in the first two weeks after the initiation of therapy might predict progression free survival (PFS) as preliminary results in literature suggest.

This is a single arm explorative phase II clinical trial in 90 subjects with advanced stage melanoma harbouring a BRAFV600 mutation. PET imaging and molecular diagnostics are combined in order to monitor response to treatment with vemurafenib plus cobimetinib, examine development of resistance and correlate changes in metabolic/proliferative activity with extend of target inhibition.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed melanoma, either unresectable stage IIIc or stage IV metastatic melanoma, as defined by AJCC 7th edition.
* Patients must be naïve to treatment for locally advanced unresectable or metastatic disease. Prior immunotherapy (including ipilimumab) is allowed.
* Documentation of BRAFV600E or BRAFV600K mutation-positive status in melanoma tumor tissue (archival or newly obtained tumor samples).
* Measurable disease per RECIST v1.1, which are accessible to biopsies.
* Biopsy lesion is within scan reach of diagnostic CT and PET-CT (thorax- abdomen-pelvis)
* ECOG performance status of 0 or 1.
* Male or female patient aged ≥ 18 years.
* Life expectancy ≥ 12 weeks.
* Adequate hematologic and end organ function within 14 days prior to first dose of study drug treatment.

Exclusion Criteria:

* History of prior RAF or MEK pathway inhibitor treatment.
* Palliative radiotherapy, major surgery or traumatic injury within 14 days prior to the first dose of study treatment.
* Active malignancy within the past 3 years other than melanoma that could potentially interfere with the interpretation of efficacy measures, except for patients with resected BCC or SCC of the skin, melanoma in-situ, carcinoma in-situ of the cervix, and carcinoma in-situ of the breast.
* History of or evidence of retinal pathology, clinically significant cardiac dysfunction, patients with active CNS lesions, renal or liver dysfunction as described in main protocol (REPOSIT NL48639.031.14).
* Pregnant, lactating, or breast-feeding.
* Unwillingness or inability to comply with study and follow-up procedures (i.e. severe anxiety disorder preventing PET/CT imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2014-12; Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Progression Free survival (PFS) | Participants will be followed until they have progressive disease based on RECIST1.1, an expected median of 10 months.
Standardized Uptake Value (SUV) of 18F-FDG and 18F-FLT as measured by PET. | Participants will be followed until they have progressive disease based on RECIST1.1, an expected median of 10 months.
RECIST 1.1 tumor size measurement on diagnostic CT. | Participants will be followed until they have progressive disease based on RECIST1.1, an expected median of 10 months.
Cut-off values of metabolic tracer uptake of 18F-FDG/FLT on PET as a measure of response. | Participants will be followed until they have progressive disease based on RECIST1.1, an expected median of 10 months.

SECONDARY OUTCOMES:
Diagnostic accuracy of metabolic tracer uptake on PET in responders and non-responders. | Participants will be followed until they have progressive disease based on RECIST1.1, an expected median of 10 months.
Glycolytic Index, Metabolic Tumor Volume and % Injected Dose of 18F-FDG/FLT on PET. | Participants will be followed until they have progressive disease based on RECIST1.1, an expected median of 10 months.
Immunohistochemical analysis of tumor tissue in responders and non-responders. | Participants will be followed until they have progressive disease based on RECIST1.1, an expected median of 10 months.
Changes of DNA in tumor tissue as measured by DNA deep sequencing analysis. | Changes from Baseline to progression, an expected median of 10 months
Changes of RNA in tumor tissue as measured by RNA expression analysis. | Changes from Baseline to progression, an expected median of 10 months
Changes of phosphoproteomic profiles in tumor tissue measured by nano-liquid chromatography coupled to tandem mass spectrometry (nanoLC-MS/MS). | Changes from Baseline to progression, an expected median of 10 months
Changes in vemurafenib and cobimetinib drug concentrations in plasma as measured by a validated Liquid Chromotography tandem Mass Spectrometry assay | Changes from Baseline to progression, an expected median of 10 months
Overall Survival (OS) | 3 years
ECOG Performance status | Participants will be followed until they have progressive disease based on RECIST1.1, an expected median of 10 months.

CONTACTS AND LOCATIONS:
Overall Officials: Fons JM Van den Eertwegh, MD PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (10):
- Netherlands (10):
  - The Netherlands Cancer Institute, Amsterdam
  - VU medical center, Amsterdam
  - Medisch Spectrum Twente, Enschede
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Maastricht University Medical Center, Maastricht
  - University Medical Center St Radboud, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - University Medical Center Utrecht, Utrecht
  - Isala Klinieken, Zwolle

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van der Hiel B, de Wit-van der Veen BJ, van den Eertwegh AJM, Vogel WV, Stokkel MPM, Lopez-Yurda M, Boellaard R, Kapiteijn EW, Hospers GAP, Aarts MJB, de Vos FYFL, Boers-Sonderen MJ, van der Veldt AAM, de Groot JWB, Haanen JBAG. Metabolic parameters on baseline and early [18F]FDG PET/CT as a predictive biomarker for resistance to BRAF/MEK inhibition in advanced cutaneous BRAFV600-mutated melanoma. EJNMMI Res. 2025 May 28;15(1):60. doi: 10.1186/s13550-025-01259-x. PMID 40434500
- [Derived] van der Hiel B, Haanen JBAG, Stokkel MPM, Peeper DS, Jimenez CR, Beijnen JH, van de Wiel BA, Boellaard R, van den Eertwegh AJM; REPOSIT study group. Vemurafenib plus cobimetinib in unresectable stage IIIc or stage IV melanoma: response monitoring and resistance prediction with positron emission tomography and tumor characteristics (REPOSIT): study protocol of a phase II, open-label, multicenter study. BMC Cancer. 2017 Sep 15;17(1):649. doi: 10.1186/s12885-017-3626-5. PMID 28915798
- See also: Site of the Netherlands Working Group on Immunotherapy of Oncology (Wino) — http://www.win-o.nl/